CLINICAL TRIAL: NCT05370534
Title: Smartphone-Based Markerless Motion Capture for Orthopaedic Clinical Use
Status: Withdrawn | Type: Observational
Why Stopped: Funding
Sponsor: University of Arkansas (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 274321; GM125503 (Other Grant/Funding Number: NIH COBRE through UArkansas)
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-02

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Motion Capture; MCA; Markers; Markerless; biomechanics
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: The investigators anticipate validating two specific actions: a box jump and walking gait. Both will be captured in two planes, coronal and sagittal. Healthy patients without musculoskeletal complaints will be voluntarily enrolled to undergo motion capture with both methods, completed during the same visit to the UAMS Human Biomechanics Laboratory.
  Each patient will perform a box jump and walking gait using each of the two modalities. We anticipate 4 hrs will be required for each patient: 1 hr for setup before the patient arrives, 1 hr for testing, and 2 hrs for data cleaning and initial processing. This work will be performed at the UAMS Human Biomechanics Laboratory (off campus on Aldersgate Road), which is equipped for this type of analysis.

SUMMARY:
The investigators propose to create a markerless smartphone-based MCA application using AR to measure joint motion and gait patterns to address this technology gap for a simple and inexpensive MCA.

DETAILED DESCRIPTION:
Aim 1 will establish a testable AR-based smartphone app that measures clinically relevant lower-extremity motion components. Existing AR code will be adapted to identify and quantify hip, knee, and ankle range of motion in both the coronal and sagittal planes. Output will be produced directly to the phone display and can also be downloadable. Both single-motion and sequential-motion (gait) measures will be captured.

Aim 2 will then compare the app-based MCA to traditional gold standard MCA in healthy volunteers. A dedicated human biomechanics lab with capability for MCA with reflective markers will be utilized to test both MCA methods. Patients will perform a box jump and normal walking gait, and the measurements from both the standard marker-based MCA system and the smartphone markerless MCA system will be statistically compared.

ELIGIBILITY:
Inclusion Criteria

* 18-65 years old
* No known spinal pathology
* No previous lower extremity surgery
* No significant cardiac history

Exclusion Criteria

* <18 or >65 years old
* Known spinal pathology
* Previous lower extremity surgery
* Significant cardiac history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be males and females between the ages of 18 years old to 65 years old that are healthy and without any active injuries limiting full participation, in particular no known spinal pathology, history of lower extremity surgery or significant cardiac history. There are no restrictions based on gender, race, or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Hip, Knee and Spine Measurements | 1 hour
  angles

CONTACTS AND LOCATIONS:
Overall Officials: David B Bumpass, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
The Principal Investigator will carefully monitor study procedures to protect the safety of research subjects and the potential for loss of confidentiality.

REFERENCES:
- [Background] Thewlis D, Waters A, Solomon LB, Perilli E. Investigating in vivo knee volumetric bone mineral density and walking gait mechanics in healthy people. Bone. 2021 Feb;143:115662. doi: 10.1016/j.bone.2020.115662. Epub 2020 Sep 25. PMID 32987197
- [Background] Kuchen DB, Eichelberger P, Baur H, Rutz E. Long-term follow-up after patellar tendon shortening for flexed knee gait in bilateral spastic cerebral palsy. Gait Posture. 2020 Sep;81:85-90. doi: 10.1016/j.gaitpost.2020.07.003. Epub 2020 Jul 6. PMID 32693350
- [Background] Kuai S, Guan X, Liu W, Ji R, Xiong J, Wang D, Zhou W. Prediction of the Spinal Musculoskeletal Loadings during Level Walking and Stair Climbing after Two Types of Simulated Interventions in Patients with Lumbar Disc Herniation. J Healthc Eng. 2019 Dec 17;2019:6406813. doi: 10.1155/2019/6406813. eCollection 2019. PMID 31929870
- [Background] Ueno R, Navacchia A, Schilaty ND, Myer GD, Hewett TE, Bates NA. Anterior Cruciate Ligament Loading Increases With Pivot-Shift Mechanism During Asymmetrical Drop Vertical Jump in Female Athletes. Orthop J Sports Med. 2021 Mar 9;9(3):2325967121989095. doi: 10.1177/2325967121989095. eCollection 2021 Mar. PMID 34235227
- [Background] Camp CL, Loushin S, Nezlek S, Fiegen AP, Christoffer D, Kaufman K. Are Wearable Sensors Valid and Reliable for Studying the Baseball Pitching Motion? An Independent Comparison With Marker-Based Motion Capture. Am J Sports Med. 2021 Sep;49(11):3094-3101. doi: 10.1177/03635465211029017. Epub 2021 Aug 2. PMID 34339317
- [Background] Di Paolo S, Zaffagnini S, Tosarelli F, Aggio F, Bragonzoni L, Grassi A, Della Villa F. A 2D qualitative movement assessment of a deceleration task detects football players with high knee joint loading. Knee Surg Sports Traumatol Arthrosc. 2021 Dec;29(12):4032-4040. doi: 10.1007/s00167-021-06709-2. Epub 2021 Sep 4. PMID 34480582
- [Background] Tsakanikas VD, Gatsios D, Dimopoulos D, Pardalis A, Pavlou M, Liston MB, Fotiadis DI. Evaluating the Performance of Balance Physiotherapy Exercises Using a Sensory Platform: The Basis for a Persuasive Balance Rehabilitation Virtual Coaching System. Front Digit Health. 2020 Nov 27;2:545885. doi: 10.3389/fdgth.2020.545885. eCollection 2020. PMID 34713032
- [Background] Paloschi D, Bravi M, Schena E, Miccinilli S, Morrone M, Sterzi S, Saccomandi P, Massaroni C. Validation and Assessment of a Posture Measurement System with Magneto-Inertial Measurement Units. Sensors (Basel). 2021 Oct 3;21(19):6610. doi: 10.3390/s21196610. PMID 34640930
- [Background] Tamura H, Tanaka R, Kawanishi H. Reliability of a markerless motion capture system to measure the trunk, hip and knee angle during walking on a flatland and a treadmill. J Biomech. 2020 Aug 26;109:109929. doi: 10.1016/j.jbiomech.2020.109929. Epub 2020 Jul 1. PMID 32807306
- [Background] Wochatz M, Tilgner N, Mueller S, Rabe S, Eichler S, John M, Voller H, Mayer F. Reliability and validity of the Kinect V2 for the assessment of lower extremity rehabilitation exercises. Gait Posture. 2019 May;70:330-335. doi: 10.1016/j.gaitpost.2019.03.020. Epub 2019 Mar 26. PMID 30947108
- [Background] Scano A, Chiavenna A, Malosio M, Molinari Tosatti L, Molteni F. Kinect V2 implementation and testing of the reaching performance scale for motor evaluation of patients with neurological impairment. Med Eng Phys. 2018 Jun;56:54-58. doi: 10.1016/j.medengphy.2018.04.005. Epub 2018 Apr 20. PMID 29681441
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Background] Walker E, Nowacki AS. Understanding equivalence and noninferiority testing. J Gen Intern Med. 2011 Feb;26(2):192-6. doi: 10.1007/s11606-010-1513-8. Epub 2010 Sep 21. PMID 20857339
- [Background] McGinley JL, Baker R, Wolfe R, Morris ME. The reliability of three-dimensional kinematic gait measurements: a systematic review. Gait Posture. 2009 Apr;29(3):360-9. doi: 10.1016/j.gaitpost.2008.09.003. Epub 2008 Nov 13. PMID 19013070
- [Background] Tanaka R, Takimoto H, Yamasaki T, Higashi A. Validity of time series kinematical data as measured by a markerless motion capture system on a flatland for gait assessment. J Biomech. 2018 Apr 11;71:281-285. doi: 10.1016/j.jbiomech.2018.01.035. Epub 2018 Feb 8. PMID 29475751